CLINICAL TRIAL: NCT05604482
Title: Detection of Disease Activity in Giant Cell Arteritis Using CXCR4-PET/CT
Brief Title: CXCR4-PET/CT for Diagnosing Giant Cell Arteritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthias Fröhlich (Other)
Responsible Party: Sponsor-Investigator, Matthias Fröhlich, Dr. med. Matthias Fröhlich, Wuerzburg University Hospital
Organization: Wuerzburg University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CXCR4_PET_CT_RZA_V2.1
Record Dates: First submitted 2022-10-30; First posted 2022-11-03 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Vasculitis; Diagnoses Disease
Keywords: Vasculitis; LV-GCA; Giant cell arteritis; FDG-PET; Imaging; CXCR4
MeSH Terms: conditions — Vasculitis; Giant Cell Arteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CXCR4-PET experimental group (Experimental): In addition to the current standard of imaging in GCA, using FDG-PET/CT, participants receive CXCR4-PET.
  Interventions: Diagnostic Test: CXCR4-PET

INTERVENTIONS:
Diagnostic Test: CXCR4-PET — New imaging modality using CXCR4 for imaging in GCA

SUMMARY:
Giant cell arteritis (GCA) is the most common vasculitis in the elderly. Accurate diagnosis is of utmost importance in order to then initiate the necessary immunosuppressive therapy. For large-vessel GCA (LV-GCA) involving the aorta and its branches, FDG-PET/CT is the standard in imaging for diagnosis and is recommended by the guidelines. However, this only indirectly visualizes inflammation through vessel wall uptake of glucose. A new PET tracer, 68Ga-pentixafor, is used to visualize the chemokine receptor CXCR4. This receptor is expressed by cells of the immune system. In the context of inflammatory processes, upregulation of CXCL12, the ligand of CXCR4, occurs in affected tissues. The chemotactic effect of this ligand leads to the immigration of CXCR4-positive inflammatory cells into the inflamed area, which can be visualized by PET using the CXCR4-specific tracer 68Ga-Pentixafor. The value of CXCR4-PET should therefore be tested in the context of LV-GCA. This study tests the benefit of CXCR4 in therapy-naïve patients with suspected LV-GCA. For this purpose, patients will receive a FDG-PET and a CXCR4-PET for direct comparison. This is an imaging-only study. Therapy will not be affected by the study. The study is single-arm and not blinded.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of GCA within 5 days of diagnosis or initiation or intensification of therapy.
* Evidence of inflammatory activity based on clinical parameters, elevated serologic markers of inflammation (CRP > 1.0 mg/dl), or a positive imaging finding on vasculitis MRI, CCDS, or FDG-PET/CT
* Ability of the patient to provide information
* Exclusion of contraindications for the performance of a PET/CT examination (see below)

Exclusion Criteria:

* Contraindications for the performance of a PET CT examination
* Pregnancy
* Allergies
* Lack of capacity of the patient to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum measurable tracer activity on 68Ga-Pentixafor PET/CT in the area of blood vessels in active GCA | 2 years
  detection of maximum measurable tracer activity on 68Ga-Pentixafor PET/CT in the area of blood vessels after a maximum of 5 days after diagnosis or when acute inflammatory activity of GCA is detected in terms of recurrence.

SECONDARY OUTCOMES:
Correlation with clinical parameters | 2 years
  Correlation of the measured tracer activity with clinically and laboratory-chemically available parameters that are collected in clinical routine. These include CRP, peripheral blood leukocyte count, calprotectin, serum amyloid A, haptoglobin and Lactate dehydrogenase and their respective progression.
Correlation with blood leukocyte count | 2 years
  Correlation of tracer uptake on imaging with CXCR4-positive peripheral blood leukocyte count.
Comparison to other imaging modalities | 2 years
  Comparison with imaging findings from vasculitis MRI imaging implemented in standard clinical practice, duplex sonography (CCDS), and, if performed as part of routine clinical practice, FDG PET/CT data.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf A Werner, MD, Study Chair — University Hospital Würzburg Oberdürrbacherstrasse 6, 97080 Würzburg, Germany,
Locations (1):
- Departement of Internal Medicine II, Rheumatology/Clinical Immunology, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frohlich M, Serfling SE, Gernert M, Guggenberger K, Higuchi T, Gerhard-Hartmann E, Weich A, Samnick S, Schmalzing M, Bley TA, Buck AK, Werner RA. Establishing C-X-C motif chemokine receptor 4 as a novel imaging target in giant cell arteritis. Arthritis Res Ther. 2026 Feb 11. doi: 10.1186/s13075-026-03747-4. Online ahead of print. PMID 41668213